CLINICAL TRIAL: NCT01145742
Title: A Collaborative Approach to Control Hypertension in Diabetes
Brief Title: Controlling Hypertension in Diabetes- Feasibility Study
Acronym: COACH-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Diane Mckee, Prof., Dept Family and Social Medicine, Albert Einstein College of Medicine
Allocation: Randomized | Model: Single Group | Purpose: Health Services Research
Other Study IDs: 2006-232
Record Dates: First submitted 2010-06-15; First posted 2010-06-17 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Type 2 Diabetes; Hypertension; Hyperlipidemia
Keywords: Type 2 diabetes; Hypertension; Health services research; Health disparities; Behavior change
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Hyperlipidemias | interventions — Home Care Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- self-management support and BP telemonitoring (Experimental): collaborative intervention involving home BP monitoring, home behavior change counseling to enhance self management, and intensification of treatment by primary care doctors
  Interventions: Behavioral: home health/primary care collaboration
- usual care (No Intervention): usual primary care management of BP. lipids, and glucose

INTERVENTIONS:
Behavioral: home health/primary care collaboration — self-management support and telemonitoring of BP and blood glucose
  Arms: self-management support and BP telemonitoring

SUMMARY:
Many primary care patients, especially in inner-city settings, do not achieve targets for blood pressure and glycemic control. There is an urgent need to enhance treatment for those who do not reach goals within the usual clinical care system. We propose to develop a multi-component intervention grounded in the Chronic Care Model, and sustainable in resource-challenged settings. Through collaboration with home health nursing and with the use of home telemetry for feedback and intensification of therapy, we will augment usual clinical services to improve health outcomes for diabetes patients who have not been able to reach therapeutic goals. There are three specific aims. First, we will establish a feasible, practical and sustainable collaborative model between the primary care sites of our practice-based research network (NYC RING), clinical researchers at the Diabetes Research and Training Center, and The Montefiore Home Health Organization, integrating the unique expertise of each of the partners and defining the roles and responsibilities of each. Second, we will develop and refine the components of the intervention, to include training primary care providers and home health nurses to integrate the technical, psychosocial and communication processes for implementation of the intervention. Third, we will assess the feasibility of the collaborative intervention by implementing the intervention for 25 primary care patients and obtain preliminary estimates of effectiveness by comparing outcomes to 25 patients receiving usual care. Our proposal includes plans to develop feasible procedures for data collection, with qualitative and quantitative methods of assessing process and outcome measures. We will use these preliminary data to revise the intervention and prepare an R18 application to further develop and test the intervention in multiple inner-city primary care sites serving low-income diabetes patients. This proposal is for secondary prevention of diabetes complications, targeting a population known for health disparities and a high burden from this chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes,
* BP above 140/90 on two health center visits,
* home touch tone phone

Exclusion Criteria:

* dementia,
* homelessness,
* language other than English or Spanish

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Blood pressure | baseline and 6 months
  Change in blood pressure, measured at partipants' homes, between baseline and 6 months

SECONDARY OUTCOMES:
Hemoglobin A1c | baseline and 6 months
  Change in A1c from baseline to 6 months
LDL Cholesterol | baseline and 6 months
  Change in LDL cholesterol from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Diane McKee, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States